CLINICAL TRIAL: NCT05789550
Title: HELICOBACTER PYLORI INFECTION IN TYPE 2 DIABETES MELLITUS IN ASSIUT UNIVERSITY HOSPITAL
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Norhan Safwat Abd El Naem Salama, doctor, Assiut University
Other Study IDs: H PYLORI Infection
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: H Pylori Infection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ALL PATIENT DIABETIC IN THIS PERIOD WILL BE INCLUDED IN THE STUDY — 1. Full clinical history with detailed history about T2DM (its duration and treatment).
  2. Full medical examination, including BMI using the formula: weight (kg)/height (m2).
  3. Laboratory investigation, including the following:
     1. Complete blood picture.
     2. Fasting blood sugar (FBS).
     3. Postprandial blood sugar (PP-BS) (2 h after 75 g glucose orally).
     4. HbA1c.
     5. Kidney function tests (serum creatinine and blood urea).
     6. Liver function tests (serum albumin, ALT, and AST).
     7. Lipid profile, which include cholesterol and triglyceride. 4)H PYLORI Ag IN Stool

SUMMARY:
The aim is to study the association of H. pylori infection with T2DM and its relation with glycated hemoglobin (HbA1c) levels

DETAILED DESCRIPTION:
Dyspepsia is a worldwide problem that affects 40% of adults. Approximately 10% of all patients presenting for endoscopy for gastrointestinal symptoms have dyspepsia [1] Helicobacter pylori is a gram-negative spiral flagellate bacillus, which normally is a resident of gastric epithelium, It can cause inflammatory cell infiltration in gastric mucosa that produces cytokines, which are not only responsible for local effects but can damage remote tissues causing extradigestive diseases like ischemic heart disease, autoimmune thyroid disease, iron deficiency anemia, idiopathic thrombocytopenic purpura, and neurologic diseases [1].

In addition to this, it is also thought to play a direct or indirect role in the pathogenesis of metabolic syndrome, non-alcoholic fatty liver disease, and type 2 diabetes [2].

Diabetes mellitus (DM) is a major public health problem, with increasing prevalence globally. The major burden (90-95%) is caused by type 2 diabetes mellitus (T2DM), which typically develops in adulthood and is characterized by variable levels of insulin resistance, impaired insulin secretion, and increased glucose production [3].

The association between DM and H. pylori infection remains controversial, although many studies have been done, which concluded that a definiterelationship exists between the two. It is hypothesized that H. pylori infection promotes atherosclerosis by altering lipid metabolism, and this leads to the metabolic syndrome, insulin resistance, and finally, to type 2 diabetes [2].

There are several lines of evidence to implicate increased susceptibility to H. pylori infection in diabetic patients. First, a diabetes-induced impairment of cellular and humoral immunity may enhance an individual's sensitivity to H. pylori infection. Second, diabetes-induced reduction of gastrointestinal motility and acid secretion may promote pathogen colonization and infection rate in the gut. Third, altered glucose metabolism may produce chemical changes in the gastric mucosa that promote H. pylori colonization [4] pylori is a gram-negative, spiral-shaped pathogenic bacterium that specifically colonizes the gastric epithelium causing chronic gastritis, peptic ulcer disease, and/or gastric malignancy [5].

H. pylori is mainly acquired in childhood by the fecaloral, oral-oral, or gastro-oral route and has been recognized as a worldwide public health problem, which is more prevalent in developing countries [6].

H. pylori infection induces an acute polymorphonuclear 7 infiltration in the gastric mucosa, which is gradually replaced by an immunologically mediated, chronic, predominantly mononuclear cellular infiltration. The mononuclear infiltration is characterized by the local production and systemic diffusion of proinflammatory cytokines that can affect remote tissues and organic [7] As a result, an increased prevalence of extradigestive diseases has been reported in those with evidence of H. pylori infection in recent years, including ischemic heart disease, autoimmune thyroid diseases, sideropenic anemia, idiopathic

thrombocytopenic purpura, neurologic diseases, and hepatobiliary diseases[8]. T2DM is an emerging pandemic, responsible for an estimated 3.8 million adult deaths worldwide [9].

The pathogenesis of T2DM is complex, with risk factors associated with lifestyle (e.g. diet, obesity, and physical activity), genetic background, and socioeconomic factors [10].

In T2DM, the pancreas can no longer produce enough insulin to overcome the cellular loss of sensitivity, resulting in the accumulation of sugar in the bloodstream [11]. Identification of treatable causes of this disease will aid in the development of strategies to delay or prevent its onset or slow its progression. Recent evidence implicates the pathological involvement of inflammation in T2DM, which is an important process induced by H. pylori infection [12]. [13], who reported that the prevalence of H. pylori infection was higher in diabetics (24%) than in controls of similar age, sex, and socioeconomical status after 3 years of follow-up, and the reinfection rate was higher in diabetic patients. [14], who reported that there was no difference in H. pylori prevalence between patient with DM and non-DM controls. [15], who reported that H. pylori infection was positively associated with HbA1c levels through a large-scale cross-sectional analysis, which indicated a role of H. pylori in impaired glucose tolerance in adults.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

- 1) Patients with T1DM. (2) Patients with age less than 35 years. (3) Patients with history of NSAIDs or alcohol intake. (4) Patients already on steroid or immunosuppressive. (5) Patients on proton pump inhibitors. (6) Patients with history of H. pylori-eradication therapy in the previous 6 months.

(7) Patients with diagnosed malignancy in previous medical records. (8) Patients with history of hematemesis. (9) Patients with severe weight loss

Ages: 35 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: cross-sectional study
Sampling Method: Non-Probability Sample
Enrollment: 146 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
The prevelance of H PYLORI Infection in type 2 DM | 11\2022 to11\2023
  The aim is to study the association of H. pylori infection with T2DM and its relation with glycated hemoglobin (HbA1c) levels

CONTACTS AND LOCATIONS:
Overall Officials: assiut Egypt, hospital, Study Chair — Egypt

REFERENCES:
- [Background] Draz U, Rathore R, Butt NF, Randhawa FA, Malik U, Waseem T. Presence of pre-diabetes in Helicobacter pylori positive versus Helicobacter pylori negative patients having dyspepsia. J Pak Med Assoc. 2018 Jun;68(6):939-941. PMID 30323363
- [Background] Haj S, Chodick G, Refaeli R, Goren S, Shalev V, Muhsen K. Associations of Helicobacter pylori infection and peptic disease with diabetic mellitus: Results from a large population-based study. PLoS One. 2017 Aug 29;12(8):e0183687. doi: 10.1371/journal.pone.0183687. eCollection 2017. PMID 28850590
- [Background] He C, Yang Z, Lu NH. Helicobacter pylori infection and diabetes: is it a myth or fact? World J Gastroenterol. 2014 Apr 28;20(16):4607-17. doi: 10.3748/wjg.v20.i16.4607. PMID 24782613
- [Background] Outlioua A, Badre W, Desterke C, Echarki Z, El Hammani N, Rabhi M, Riyad M, Karkouri M, Arnoult D, Khalil A, Akarid K. Gastric IL-1beta, IL-8, and IL-17A expression in Moroccan patients infected with Helicobacter pylori may be a predictive signature of severe pathological stages. Cytokine. 2020 Feb;126:154893. doi: 10.1016/j.cyto.2019.154893. Epub 2019 Dec 24. PMID 31877554
- [Background] Malaty HM. Epidemiology of Helicobacter pylori infection. Best Pract Res Clin Gastroenterol. 2007;21(2):205-14. doi: 10.1016/j.bpg.2006.10.005. PMID 17382273
- [Background] Eskandarian R, Ghorbani R, Shiyasi M, Momeni B, Hajifathalian K, Madani M. Prognostic role of Helicobacter pylori infection in acute coronary syndrome: a prospective cohort study. Cardiovasc J Afr. 2012 Apr;23(3):131-5. doi: 10.5830/CVJA-2011-016. PMID 22555636
- [Background] Mishra RR, Tewari M, Shukla HS. Association of Helicobacter pylori infection with inflammatory cytokine expression in patients with gallbladder cancer. Indian J Gastroenterol. 2013 Jul;32(4):232-5. doi: 10.1007/s12664-013-0321-6. Epub 2013 Feb 28. PMID 23446740
- [Background] van Dieren S, Beulens JW, van der Schouw YT, Grobbee DE, Neal B. The global burden of diabetes and its complications: an emerging pandemic. Eur J Cardiovasc Prev Rehabil. 2010 May;17 Suppl 1:S3-8. doi: 10.1097/01.hjr.0000368191.86614.5a. PMID 20489418
- [Background] Agardh E, Allebeck P, Hallqvist J, Moradi T, Sidorchuk A. Type 2 diabetes incidence and socio-economic position: a systematic review and meta-analysis. Int J Epidemiol. 2011 Jun;40(3):804-18. doi: 10.1093/ije/dyr029. Epub 2011 Feb 19. PMID 21335614
- [Background] Papamichael KX, Papaioannou G, Karga H, Roussos A, Mantzaris GJ. Helicobacter pylori infection and endocrine disorders: is there a link? World J Gastroenterol. 2009 Jun 14;15(22):2701-7. doi: 10.3748/wjg.15.2701. PMID 19522019